CLINICAL TRIAL: NCT01604200
Title: A Mixed Methods Study to Assess How to Engage Dentists in Blood Pressure Screening
Brief Title: Dental PROBE (Dental Practice suRvey of Office Blood Pressure mEasurement)
Acronym: Dental-PROBE
Status: Withdrawn | Type: Observational
Why Stopped: Funding unsuccessful
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Sheldon Tobe, Associate Professor Department of Medicine, University of Toronto, Sunnybrook Health Sciences Centre
Other Study IDs: 292-2011
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Focus of Study is on Dentist's Attitudes Toward BP Measures
Keywords: hypertension; dentistry; blood pressure; measurement; screening; qualitative research
MeSH Terms: conditions — Hypertension | interventions — Focus Groups

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dentists: Dentists in practice
  Interventions: Behavioral: focus group

INTERVENTIONS:
Behavioral: focus group — key informant review

SUMMARY:
20% of Canadians are hypertensive with approximately 200,000 new cases each year. Early detection of hypertension affects outcomes, reducing the risk for heart attack, stroke, kidney disease, and dementia. Screening strategies are required to identify the more than one third of Canadians with unrolled high blood pressure, in particular, younger men unaware of their condition, women over sixty years old, and underserved groups.

A collaborative practice model linking dentists to other healthcare providers in a reporting network is a promising model for hypertension detection and management. There are 20,129 licensed dentists in Canada who graduate with the ability to measure blood pressure, and 74% of the population visits a dentist each year. This represents an opportunity, but information is required on Dental attitudes toward screening for hypertension before attempting to initiate a screening model. To engage dentists in hypertension detection requires an understanding of the practice environment and the factors that shape their beliefs, attitudes and behaviours regarding routine hypertension screening in their practices.

ELIGIBILITY:
Inclusion Criteria:

* Dentists in practice

Exclusion Criteria:

* Unwilling to participate in study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Canadian dental faculties and regulators. Canadian dentists. Canadian dental patients. Canadian dental experts
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada